CLINICAL TRIAL: NCT06052488
Title: Strength After Breast Cancer: Clinical Implementation of an Evidence-based Group Exercise Intervention for Breast Cancer Survivors
Brief Title: Strength After Breast Cancer
Acronym: SABC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Responsible Party: Principal Investigator, Stephen Wechsler, Principal Investigator, MGH Institute of Health Professions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-418
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Physical Therapy; Exercise Program
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strength After Breast Cancer (SABC) Intervention (Experimental): Participants will undergo study procedures as outlined:
  * Complete a baseline survey regarding exercise self-efficacy, physical activity level, quality of life, and fatigue
  * Attend a 1-on-1 physical therapy evaluation and 4 group exercise sessions at MGH Waltham
  * After completing the 4 exercise sessions, complete follow-up surveys including a program satisfaction survey
  * At 1-month post-program, complete follow-up surveys and an individual, semi-structured interview with study staff to supply feedback about the program.
  * At 3-months post-program, complete follow-up surveys
  Interventions: Behavioral: Strength After Breast Cancer

INTERVENTIONS:
Behavioral: Strength After Breast Cancer — Individual physical therapy evaluation and 4 group-based exercise sessions led by a licensed physical therapist

SUMMARY:
The goal of this study is to explore whether a group exercise program called Strength After Breast Cancer can be delivered in an outpatient physical therapy clinic to improve physical function among women after treatment for breast cancer.

The main questions this study aims to answer are:

* Can the Strength After Breast Cancer program and the associated outcome battery be successfully delivered in an outpatient physical therapy clinic at Massachusetts General Hospital and do participants find the program practical?
* What are the barriers to and facilitators of delivering the group exercise program in a clinical setting and what changes need to be made to the program to improve sustainability and to facilitate implementation at other clinical sites?

Participants will complete study questionnaires before and after engaging in the group exercise program and they will participate in interviews following participation in the program.

DETAILED DESCRIPTION:
The goal of this single arm feasibility study of the Strength After Breast Cancer (SABC) evidence-based group exercise intervention for women after treatment for breast cancer is to determine if investigators can feasibly deliver the program out of the outpatient physical therapy clinic at Massachusetts General Hospital Waltham.

- Following a one-on-one physical therapy evaluation, the four-session SABC program provides a group-based but individualized exercise plan and encourages engagement in independent home-based exercises to improve physical function. The SABC program has previously been found to be safe and led to improvements in physical function among women after treatment for breast cancer. Therefore, the focus of this study is to explore clinical implementation barriers, facilitators, and necessary program adaptations to enhance sustainability and facilitate implementation at other clinical sites.

Study procedures include screening for eligibility, in-clinic visits, questionnaires, and a semi-structured interview.

Participation in this research study is expected to last up to 5 months. It is expected that up to 40 people will take part in this research study.

This is an unfunded study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosed with Stage I-III breast cancer, having completed primary cancer treatment (e.g., surgery, chemotherapy, radiation therapy); hormonal therapies and adjuvant targeted therapies will be permitted

Exclusion Criteria:

* Any injury or medical condition that would prohibit being able to safely perform exercise as indicated by the Physical Activity Readiness Questionnaire (i.e., atrial fibrillation, chest pain or angina, uncontrolled high blood pressure or hypertension, loss of balance due to dizziness in the past 12 months, or loss of consciousness in the past 12 months).
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — These eligibility criteria are aligned with the criteria outlined by the developers of the Strength After Breast Cancer program. This program was developed for women after treatment for breast cancer.
Enrollment: 40 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Screening Rate | At screening
  Number patients screened / Number patients identified as potentially eligible. Screening rate of at least 75% will indicate feasibility.
Eligibility Rate | At screening
  Number patients screening eligible / Number screened. Eligibility rate of at least 75% will indicate feasibility.
Enrollment Rate | At screening
  Number participants enrolled / Number screened positive & eligible. A rate of at least 75% will indicate feasibility.
Program completion rate | Up to 2 months
  Number participants completing 4 sessions of the SABC intervention / Number of participants enrolled. For this study, the investigators will consider it feasible if 75% of participants complete all 4 sessions.
Intervention session completion rate | Up to 2 months
  Number of completed sessions per participant. For this study, the investigators will consider it feasible if the mean number of sessions completed per participant is ≥ 3.
Assessment completion rate | Up to 5 months
  Number participants completing each of the 4 study assessments / Number of participants enrolled. For this study, an assessment completion rate of 75% will indicate feasibility.

SECONDARY OUTCOMES:
Participant Satisfaction | Up to 2 months
  Assessed by the post-program satisfaction survey which is a 7-item survey that is rated on a 5-point Likert scale; total score range 7-35 (higher score indicates greater satisfaction). Any item on the Satisfaction survey that generates a mean score of < 4 will trigger consideration of modification to the SABC program.
Exercise Self-Efficacy | Up to 5 months
  Assessed with the Self-Efficacy with Exercise scale which consists of nine potential exercise barriers and asks the individual to rate their confidence on a 0 (not confident) - 10 (very confident) scale that they could exercise for twenty minutes, three times per week, given each barrier (total score range 0-90; maximum score of 90 indicates highest exercise self-efficacy).
Physical Activity Level | Up to 5 months
  Assessed using the International Physical Activity Questionnaire Long Form to assess duration and frequency of physical activity in the last seven days in domains of: job-related, transportation, housework/house maintenance/caring for family, recreation/sport/leisure-time, and time spent sitting.
Quality of Life: Functional Assessment of Cancer Therapy - General | Up to 5 months
  Assessed using the Functional Assessment of Cancer Therapy - General (FACT-G) (28 items), which measures health-related quality of life covering four domains of well-being (physical, social/family, emotional, functional). This measure is included in and will be assessed as part of The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F). Total score range for FACT-G is 0-108 with higher scores indicating greater quality of life.
Cancer-Related Fatigue: Functional Assessment of Chronic Illness Treatment - Fatigue, Fatigue subscale | Up to 5 months
  Assessed using the Functional Assessment of Chronic Illness Treatment - Fatigue (FACIT-F), 13 item fatigue subscale. Total score for 13-item fatigue subscale is 0-52 with higher score indicating worse fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wechsler, DPT, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- MGH Institute of Health Professions, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: the Partners Innovations team at http://www.partners.org/innovation. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation